CLINICAL TRIAL: NCT05237505
Title: The Cardiovascular Consequences of Sleep Apnea Plus COPD (Overlap Syndrome)
Acronym: CRESCENDO-SLP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Atul Malhotra, Professor, Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 808025
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea; Chronic Obstructive Pulmonary Disease; Overlap Syndrome
Keywords: OSA; obstructive sleep apnea; COPD; chronic obstructive pulmonary disease; PAP therapy; oxygen; cardiovascular health
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation; nitrox

STUDY DESIGN:
Intervention Model Description: 6-month, 2-arm randomized, parallel, interventional mechanistic study of COPD/OSA overlap syndrome to compare bi-level PAP vs. O2 therapy
  Qualified participants will be randomized to receive either O2 therapy or bi-level therapy.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen (Experimental): OVS subjects will receive treatment with oxygen during night time for 6 months
  Interventions: Drug: Oxygen gas
- Bi-level positive pressure non invasive ventilation (Experimental): OVS subjects will receive treatment with bi-level PAP therapy during night time for 6 months
  Interventions: Device: bi-level positive pressure non invasive ventilation

INTERVENTIONS:
Device: bi-level positive pressure non invasive ventilation — Participants randomized to the bi-level arm will be provided with an auto bi-level device that automatically delivers the required pressure. The settings in the auto bi-level will be minimum EPAP of 4 cmH2O, maximum IPAP of 24 cmH2O, and a range of pressure support between 6-10 cmH2O. For those participants who have been randomized to the bi-level group but have not successfully acclimated to the device with the automatic bi-level settings, we will conduct an in-lab titration of the bi-level therapy during the optional Overnight visit 2.
  Other Names: Auto-bilevel; BIPAP; Non invasive ventilation
  Arms: Bi-level positive pressure non invasive ventilation
Drug: Oxygen gas — The dose of nocturnal oxygen in all participants in the oxygen therapy arm will be 2 liters/minute. Patients with daytime hypoxemia, measured as sustained desaturations below 89% during wake time and/or arterial blood PO2 ≤ 55 mmHg, will be excluded from this study (as specified in the exclusion criteria) for ethical reasons since withholding oxygen in hypoxemic patients would be at odds with standard of care.
  Other Names: O2
  Arms: Oxygen

SUMMARY:
Major progress has been made in the area of cardiovascular disease, but we believe that further progress will involve mechanistically addressing underlying respiratory causes including chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea (OSA). The most common cause of death in COPD is cardiovascular, although mechanisms are unknown. OSA has been associated with major neurocognitive and cardiovascular sequelae, the latter likely a function of autonomic nervous system abnormalities, oxidative stress, inflammation, and other pathways. Recent data suggest that individuals with OVS die preferentially of cardiovascular disease compared to OSA or COPD alone, although mechanisms are again unclear.

The combination of OSA and COPD may lead to profound hypoxemia. Individuals with COPD can develop pulmonary hypertension via disturbances in gas exchange and parenchymal injury leading to loss of pulmonary vasculature. OSA has been associated with mild to moderate pulmonary hypertension, but the situation may be worse if combined with parenchymal lung disease. The biological response to sustained hypoxemia has been carefully studied as has the topic of intermittent hypoxemia; however, to our knowledge, very little research has occurred regarding the combination of sustained plus intermittent hypoxia as seen in OVS. For example, we do not really know whether individuals with OVS develop coronary disease, right or left heart failure, dysrhythmias or some combination of abnormalities predisposing them to cardiovascular death. Thus, design of interventional studies is challenging as causal pathways are poorly understood despite our considerable preliminary data addressing these issues.

The purpose of this study is to examine vascular mechanisms in individuals with COPD/OSA overlap syndrome (OVS) compared with matched individuals with obstructive sleep apnea (OSA) alone or chronic obstructive pulmonary disease (COPD) alone and to perform a phase II pilot mechanistic clinical trial in OVS to examine the effect size of nocturnal bi-level positive airway pressure (PAP) vs. nocturnal oxygen therapy in cardiovascular outcomes.

DETAILED DESCRIPTION:
For Aim 1, we will perform a cross-sectional clinical study that will allow us to test the hypothesis that individuals with OVS have increased markers of vascular risk compared with matched individuals with OSA alone or COPD alone. This aim will also allow us to compare the magnitude of the effect of OSA vs. COPD vs OVS for design of subsequent basic and clinical studies.

For Aim 2, we will perform a randomized 1:1 clinical trial stratified by sex that will allow us to test the hypothesis that bi-level PAP therapy is superior to oxygen in the treatment of individuals with OVS from the standpoint of right ventricular mass (primary outcome) and other cardiovascular risk parameters/outcomes. We will use these interventions as tools to explore their impacts on important biomarkers of interest e.g., miR210 may predict risk of atherosclerosis and changes in levels may give insight into mechanisms of our interventions. There is no sub-study analysis. The aim of the interventional section of this study (aim 2) is to analyze the effect on cardiovascular outcomes of both nocturnal oxygen therapy and bi-level therapy on patients with COPD-OSA overlap syndrome.

Participants will undergo the following activities:

* Eligibility screening (online or via phone; ~10 minutes)
* Subjects who screen positive: In-person eligibility assessment (~1.5 hours) including a history, exam, questionnaires, spirometry, and an overnight home sleep test.
* Participants who are eligible: Will come to the research lab for an overnight visit (~12 hours) which includes the following activities: general exam, questionnaires, blood test, measures of cardiovascular health (e.g., blood pressure), neurocognitive function (e.g., a memory test), a pulmonary function test, and an overnight sleep study to assess the severity of sleep apnea.
* After overnight visit 1, participants will come to day time visit 2 for the cardiac MRI. After this visit, participants who are only COPD or only OSA will have completed the study. Participants with OVS will be offered to continue the study. Participants will come to the research lab for a mask adaptation day visit; if they can tolerate a bilevel mask, they will be randomized to the oxygen versus the bi-level arm. We will ask participants to be on the therapy for 6 months, during which time the research team will make weekly calls to check adherence to the therapies.
* After 6 months on the treatment, OVS participants will come back to an overnight visit which includes the following tests: general exam, questionnaires, blood test, measures of cardiovascular health (e.g., blood pressure), neurocognitive function (e.g., a memory test), and an overnight sleep study. Additionally, they will have a day time visit for the Cardiac MRI.

Researchers will compare the effects of bi-level PAP on cardiovascular health with the effects of oxygen to see if bi-level may be an effective treatment for select patients with OVS.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Persons aged 40-79.
* For women, only postmenopausal women will be included
* Diagnosed with untreated moderate to severe obstructive sleep apnea (apnea-hypopnea index ≥15 events/hr and ≤80 events/hr) and/or diagnosed with COPD with FEV1/FVC ratio <0.7 and will be on stable medications as assessed by a board-certified pulmonologist.

Exclusion Criteria:

* Premenopausal women (i.e. women are pregnant or may become pregnant) or lactation
* Presence of specific devices: cardiac implantable electronic device (CIED) such as pacemakers, implantable cardioverter defibrillators (ICDs) and cardiac resynchronization therapy (CRT) devices, metallic foreign bodies, implantable neurostimulation systems, cochlear implants/ear implant, drug infusion pumps (insulin delivery, analgesic drugs, or chemotherapy pumps), metallic fragments such as bullets, shotgun pellets, and metal shrapnel , cerebral artery aneurysm clips, magnetic dental implants, and artificial limb.
* Known allergic reactions to components of the study intervention: (if getting contrast, MRI contrast (gadolinium)).
* Concurrent severe sleep disorders (such as periodic limb movements, restless legs syndrome, narcolepsy, idiopathic hypersomnia, etc).
* Exhibit Cheyne-Stokes respiration or central sleep apnea (> 25 % of events central)
* Take potentially confounding medications or hormones that affect breathing.
* Subjects will be excluded if they are deemed medically unstable with active neurological, cardiac, liver, endocrine, and infectious diseases.
* We will also exclude participants with pulmonary disease apart from COPD.
* We will exclude participants with active cancer treatment.
* We will exclude azotemia (estimated glomerular fraction rate < 30ml/min) as there is some concern about giving gadolinium to these patients (if getting contrast MRI).
* people with exposures deemed to be problematic for the research e.g. any smoking in bedroom by participant or household member, major second-hand smoke, e-cigarettes, tetrahydrocannabinol, major drug or alcohol consumption (>3 oz/day) and other environmental pollution effects (indoor and outdoor).
* Individuals who are already on continuous O2 for COPD or PAP treatment for OSA.
* Patients with sustained desaturations below 89% during wake time will be excluded for ethical reasons since withholding oxygen in hypoxemic patients would be at odds with standard of care.
* Individuals with OSA (AHI range 15-80/hr) will be screened for pathological sleepiness and will be excluded if ESS >18/24, history of motor vehicle accident or near miss accident, or high-risk occupation.
* COPD individuals with arterial PCO2 higher than 52 mmHg will be excluded.
* Individuals who are currently incarcerated.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Right ventricular mass | 6 Months
  Cardiac magnet resonance imaging (CMRI): All subjects will undergo cardiac MRI measurements the same day they undergo the evaluation of vascular reactivity measurements. Supine cardiac MRI imaging will be performed using a 3T MR scanner (GE 750, GE Healthcare) with a 16-element cardiac coil for radiofrequency signal reception. Non-invasive blood pressure will be monitored during cardiac MRI scanning (Dinemap). Standard and novel MRI sequences will be used for myocardial tissue characterization, assessment of ventricular function, pulmonary hemodynamics, and aortic compliance
Reactive Hyperemia Index | 6 months
  Based on a device called EndoPAT, which measures non-invasively bloodflow before, during, and after 5-minutes of occlusion to one arm.
5th generation troponin | 6 months
  Troponin will be measured from participant serum samples. Troponin is a marker of myocardial injury.
MiR-210 | 6 months
  MicroRNA-210 will be measured from participant serum samples. miR210 may predict risk of atherosclerosis and changes in levels may give insight into mechanisms of our interventions

SECONDARY OUTCOMES:
Verbal Paired-Associates task | 6 months
  Participants will complete a word pairs task, which is a computerized memory assessment designed to prime participants to memorize 26 pairs of words in the evening. To assess sleep-dependent memory consolidation, recall of these word pairs are tested in the morning after the overnight sleep study.
Response Speed | 6 months
  Objective assessment of brain function will be done using 10-minute psychomotor vigilance test

CONTACTS AND LOCATIONS:
Overall Officials: Atul Malhotra, MD, Principal Investigator — UCSD
Locations (1):
- UCSD Sleep Research, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No